CLINICAL TRIAL: NCT02848222
Title: Pilot Study for Investigating the Effect of the Bruder Eye Hydrating Compress on Contact Lens Discomfort in Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Bruder Healthcare Company (Unknown)
Responsible Party: Principal Investigator, Jason Nichols, principal investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR1016
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Contact Lens Discomfort; Dry Eye Disease; Meibomian Gland Dysfunction
Keywords: contact lens discomfort; dry eye disease; meibomian gland dysfunction; Bruder mask
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

ARMS (3):
- Twice Daily Application of Bruder compress (Experimental): Ten minute application of the Bruder Moist Heat Compress in the morning prior to contact lens insertion and ten minute application in the evening after lens removal
  Interventions: Device: Bruder Moist Heat Compress
- Once Daily Application of Bruder compress (Experimental): Ten minute application of the Bruder Moist Heat Compress in the evening after lens removal
  Interventions: Device: Bruder Moist Heat Compress
- Twice Daily Application of warm washcloth (Sham Comparator): Ten minute application of a hot-water warmed washcloth in the morning prior to contact lens insertion and ten minute application in the evening after lens removal
  Interventions: Other: Washcloth

INTERVENTIONS:
Device: Bruder Moist Heat Compress
  Other Names: Bruder mask
  Arms: Once Daily Application of Bruder compress; Twice Daily Application of Bruder compress
Other: Washcloth
  Arms: Twice Daily Application of warm washcloth

SUMMARY:
The purpose of this prospective study is to evaluate the benefits of using the Bruder Moist Heat Compress in contact lens wearers who report reduced comfortable wear time. This will be done by assessing for improvement in ocular oil gland function and comfortable contact lens wearing time after one month of daily warm compress application. The efficacy of the Bruder Moist Heat Compress applied once will be compared to twice daily application as well as compared to warm compress application using a wash cloth.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Provide informed consent and authorization to disclose protected health information
* Have habitual contact lens corrected visual acuity in each eye of at least 20/30
* Willing to comply with protocol
* Wear soft daily contact lenses for total wear time of at least 4 hours a day and at least 4 days a week on average over at least a 30 day period before enrollment

Exclusion Criteria:

* Have any uncontrolled systemic disease that in the investigator's opinion could be expected to interfere with the study, for example, conditions associated with dry eye disease
* Pregnant by self-report
* Active ocular conditions: infection, allergic conjunctivitis, severe eyelid inflammation including anterior blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Twice Daily Application of Bruder Compress: Ten minute application of the Bruder Moist Heat Compress in the morning prior to contact lens insertion and ten minute application in the evening after lens removal
- Group 2: Once Daily Application of Bruder Compress: Ten minute application of the Bruder Moist Heat Compress in the evening after lens removal
- Group 3: Twice Daily Application of Warm Washcloth: Ten minute application of a hot-water warmed washcloth in the morning prior to contact lens insertion and ten minute application in the evening after lens removal
Period: Overall Study
Arm/Group | Group 1: Twice Daily Application of Bruder Compress | Group 2: Once Daily Application of Bruder Compress | Group 3: Twice Daily Application of Warm Washcloth
Started | 25 | 18 | 17
Completed | 18 | 17 | 17
Not Completed | 7 | 1 | 0

BASELINE CHARACTERISTICS:
Population: While 18 subjects in Group 1 completed all visits in the study, one subject's data was not used in the analysis due to poor compliance with instructions on using the Bruder compress and inaccessibility to an appropriate heating appliance for a prolonged period of time during the study period. Thus, only 17 subjects' data were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Twice Daily Application of Bruder Compress | Group 2: Once Daily Application of Bruder Compress | Group 3: Twice Daily Application of Warm Washcloth | Total
Number analyzed (Participants) | 17 | 17 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (8) | 32 (12) | 36 (11) | 33 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 17 | 50
  Male | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 1 | 2 | 5
  Race: Native Hawaiian or Pacific Islander | 0 | 2 | 0 | 2
  Race: Caucasian | 10 | 8 | 8 | 26
  Race: African American | 5 | 6 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 17 | 51
Comfortable Contact Lens Wear Time [Mean (Standard Deviation); unit: hours per day] | 7.8 (3.0) | 8.0 (3.9) | 5.9 (3.2) | 7.3 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Duration of Subject-reported Comfortable Contact Lens Daily Wear Time (Hours Per Day)
Time Frame: Baseline through 1 month
Population: In Gr1, 25 subjects were randomized, 18 subjects completed, 7 discontinued early and 1 subject's data was not used due to poor compliance resulting in 17 subjects analyzed. In Gr2, 18 subjects were randomized and 17 completed. In Gr3, 17 subjects were randomized and completed.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Group 1: Twice Daily Application of Bruder Compress | Group 2: Once Daily Application of Bruder Compress | Group 3: Twice Daily Application of Warm Washcloth
Number analyzed (Participants) | 17 | 17 | 17
hours per day | 9.2 (2.8) | 8.5 (3.6) | 7.1 (2.8)
Statistical Analysis 1: Comparison: Group 1: Twice Daily Application of Bruder Compress vs Group 2: Once Daily Application of Bruder Compress vs Group 3: Twice Daily Application of Warm Washcloth; Test type: Superiority; p = 0.02, ANOVA — Threshold for significance was p < 0.05

ADVERSE EVENTS:
Time Frame: Baseline through 1 month
Arm/Group | Group 1: Twice Daily Application of Bruder Compress | Group 2: Once Daily Application of Bruder Compress | Group 3: Twice Daily Application of Warm Washcloth
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/25 | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT02848222/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT02848222/SAP_001.pdf